CLINICAL TRIAL: NCT00938990
Title: The Effect of Etomidate on Outcomes of Trauma Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Advocate Hospital System (Other)
Responsible Party: Principal Investigator, Erik Kulstad, MD, MS, Research Director, Advocate Hospital System
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4667 - ACH IRB
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Etomidate; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam
- Etomidate (Experimental)
  Interventions: Drug: Etomidate

INTERVENTIONS:
Drug: Etomidate
  Arms: Etomidate
Drug: Midazolam
  Arms: Midazolam

SUMMARY:
Rationale: The drug etomidate causes increased mortality if used for continuous sedation in mechanically ventilated patients; however, etomidate continues to be widely used as a single-bolus induction agent for endotracheal intubation because of its favorable hemodynamic properties. Recent data have raised questions regarding the safety of using etomidate for even a single bolus in patients at risk of adrenal insufficiency, emphasizing the fact that single bolus doses of etomidate cause measurable adrenal suppression, and consequently may cause increases in vasopressor requirements and in hospital length of stay. Alternative FDA-approved induction agents, such as midazolam, may be safer than etomidate; however, no studies have formally compared these agents.

Research Hypothesis: The investigators hypothesize that in critically ill trauma patients presenting to the emergency department requiring rapid sequence intubation, the hospital length of stay for patients given etomidate will be greater than for patients given midazolam for induction.

Specific Aims: The specific aim is to determine the difference in hospital length of stay between trauma patients given etomidate and those given midazolam for induction during rapid sequence intubation in the emergency department. The investigators plan to compare the two groups in terms of hospital length of hospital stay, length of stay in the intensive care unit, and duration of intubation by performing a prospective, randomized, trial of critically ill trauma patients presenting to the emergency department requiring intubation. The investigators will also compare the mortality rates in these two groups while controlling for severity of illness and the use of steroids while hospitalized.

Significance: If the use of etomidate to induce anesthesia prior to intubation adversely affects the hospital length of stay of trauma patients, this length of stay might be reduced in such patients by using alternative agents for induction. Since etomidate is currently in widespread use as an induction agent, the results of this study could have significant implications for patient management.

ELIGIBILITY:
Inclusion Criteria:

* All critically ill trauma patients (defined as patients over the age of 14 years requiring trauma team activation) who present to the ED in need of ventilatory support due to the severity of their illness and injuries.

Exclusion Criteria:

* Age less than 14, do-not-resuscitate status, or cardiopulmonary arrest prior to arrival in the ED.

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Length of Stay